CLINICAL TRIAL: NCT02146196
Title: Roboter-unterstützte Kardiale Rehabilitation Herzinsuffzienter Patientinnen Und Patienten
Brief Title: Robotic Assisted Rehabilitation for Heart Failure Patients and Patients After Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZH_2011_0119
Record Dates: First submitted 2014-05-11; First posted 2014-05-23 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Heart Failure; Post Cardiac Surgery
Keywords: Heart failure; robotic assisted gait therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heart failure, robotic assisted training (Experimental): 4 weeks robotic assisted training with the Lokomat®
  Interventions: Device: 4 weeks robotic assisted training with the Lokomat®
- Post cardiac surgery (Experimental): One week robotic assisted gait training with the Lokomat®
  Interventions: Device: One week robotic assisted gait training with the Lokomat®

INTERVENTIONS:
Device: 4 weeks robotic assisted training with the Lokomat® — During a prespecified time period (4weeks) a three times weekly robotic assisted gait training during 30-45 minutes. Strength training, interval training and endurance training are possible.
  Arms: Heart failure, robotic assisted training
Device: One week robotic assisted gait training with the Lokomat® — During a prespecified time period (1week) a three times weekly robotic assisted gait training during 10-40 minutes. Strength training, interval training and endurance training are possible
  Arms: Post cardiac surgery

SUMMARY:
Robotic assisted gait therapy with the Lokomat® as a new method for rehabilitation in advanced heart failure and after cardiac surgery.

DETAILED DESCRIPTION:
Rehabilitation in heart failure medicine is limited due to many comorbidities and reduced exercise capacity in this patient group. In patients after cardiac surgery rehabilitation is sometimes difficult especially due to ICU- acquired weakness following a prolonged intensive care course. To tackle these problems and enable recovery and rehabilitation many of the conventional methods are lacking feasibility. During the next decades increasing numbers of older and more frail patients in the field of advanced heart failure are expected. To establish a new method for rehabilitation we use technology well established in other divisions of medicine. Robotic assisted gait therapy is well established in neurology in paraplegic and tetraplegic patients, patients after stroke and traumatic injured patients. Gait therapy is used to re-establish the normal course of motion. The Lokomat ® (Hocoma AG) is therefore used in over 25 countries worldwide. The combination of different training modes (interval training, endurance training and resistance training) is one of the advantages. The most important benefit is the possibility to extend or relieve the robotic assistance up to a point without support on the one hand and full support from the Lokomat ® on the other hand and relieve the patient partly or complete from his bodyweight. This enables the therapist to plan the most possible individual training almost independent from his exercise capacity for each patient. Up to now heart failure is a contraindication for training with the Lokomat ® and no trial was performed after cardiac surgery. Therefore a clinical trial is necessary to establish this method in the field of heart failure medicine and after cardiac surgery. In our prospective trial we investigate two points after a feasibility trial first, were healthy persons and patients with NYHA 1 or less are trained for safety reasons, to establish possible protocols and get familiar with the robotic assisted gait therapy. In the prospective trial we train patients with stable heart failure (NYHA 2 or NYHA 3) and a left ventricular ejection fraction less than 45% for 4 weeks with 3 trainings per week.

Timeframe for heart failure Patients: Screening day0; Baseline/Start of the training day0 +(0-5days); training period day0+ (0-5days) up to 4 Weeks, 28 days of training with the Lokomat®. Each week three training periods; End of Study Visit after 4 to 5 Weeks from baseline.

Timeframe for patients after cardiac surgery: Screening day0; baseline/start of the training day0 +(0-2days); training period one week with the Lokomat® with three training sessions; end of study visit after one week, telephone follow up twelve weeks after hospital discharge to evaluate possible deep sterna wound infection. Due to the character as a pilot trial, there are no statistical end points, but stress test (spiroergometry), blood sample (interleukin 6, CRP, BNP) , strength measurement of the Musc. quadriceps and a quality of life questionnaire (SF 36) are taken at baseline (day0) and after the 4 week training period at end of study visit. Patients after cardiac surgery are trained with another strategy. There the safety aspect is the most important in this pilot trial. Patients after cardiac surgery are trained with the Lokomat® during initial hospitalization for one week with three sessions. A six minute walk test and measurement of quadriceps peak force is done at at baseline/start of the training day0, expected at day 3 to 14 after surgery, and after one week of training at end of study visit day seven. A telephone follow up of this patients three months after hospital discharge is done for possible deep sternal wound infection.

Each training in the heart failure group should lasts 30-45minutes. The heart failure group should contain 5-6 patients. The training in the postcardiotomy group should last 10-40minutes depending on patients postoperative status. The postcardiotomy group should contain 10 patients. 20 patients receiving normal postoperative physiotherapy serve as a control group.

ELIGIBILITY:
Inclusion Criteria:

Heart failure patients:

* stable heart failure (over 3 months, NYHA 2, NYHA 3)
* Left ventricular ejection fraction less than 45% postoperative patients:
* possibility to walk at least 50m on the ground floor

Exclusion Criteria:

* weight >100kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Deep sternal wound infections | 12 weeks after hospital discharge
  Occurence of deep sternal wound infections due to training, only in patients after cardiac surgery
Changes in VO2 (maximal oxygen uptak in ml/(kg*min)) | After four weeks robot-assisted training with the Lokomat®
  Change in maximal oxygen uptake during spiroergometry due to training, only in heart failure patients
Changes in BNP | After four weeks robot-assisted training with the Lokomat®
  Change in brain natriuretic peptide due to training, measured in mg/ml. Only in heart failure patients.
Changes in strength measurement of the musculus quadriceps | After four weeks robotic assisted training with the Lokomat®. In the postcardiotomy group after one week robot-assisted training
  isometric strength of the musculus quadriceps measured in kilopond
Changes in CRP (C- reactive protein) | After four weeks robot-assisted training with the Lokomat®
  Change in C- reactive protein, due to training, measured in mg/ml. Only in heart failure patients.
Changes in IL 6 (interleukin 6) | After four weeks robot-assisted training with the Lokomat®
  Change in interleukin 6(measured in mg/ml), due to training. Only in heart failure patients.
Changes in SF 36 | After four weeks robot-assisted training with the Lokomat®
  Questionaire (SF 36- short form 36 of health survey) to assess changes in quality of life due to the training. Only in heart failure patients
Changes in walking distance (in meters) in 6 minute walk test (MWT) | After one week robot-assisted training with the Lokomat®
  6 minute walk test to assess changes in walking distance after training period, only in patients after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Volkmar Falk, MD, Study Director — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Schoenrath F, Markendorf S, Brauchlin AE, Frank M, Wilhelm MJ, Saleh L, Riener R, Schmied CM, Falk V. Robot-assisted training for heart failure patients - a small pilot study. Acta Cardiol. 2015 Dec;70(6):665-71. doi: 10.2143/AC.70.6.3120178. PMID 26717214
- [Derived] Schoenrath F, Markendorf S, Brauchlin AE, Seifert B, Wilhelm MJ, Czerny M, Riener R, Falk V, Schmied CM. Robot-Assisted Training Early After Cardiac Surgery. J Card Surg. 2015 Jul;30(7):574-80. doi: 10.1111/jocs.12576. Epub 2015 May 22. PMID 25998717